CLINICAL TRIAL: NCT00890006
Title: Low-Intermediate Risk Prostate Cancer: Improving Acute Toxicity Outcomes of Radiotherapy With the Integration of Advanced Imaging for Treatment Planning and Guidance
Brief Title: Advanced Imaging for Radiotherapy Treatment Planning and Guidance for Low-Intermediate Risk Prostate Cancer (Margin)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 06-0520-C
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Low or Intermediate Risk Prostate Cancer
Keywords: Prostate cancer; Magnetic resonance imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI + CBCT in prostate cancer (Experimental)
  Interventions: Procedure: Advanced imaging for radiotherapy planning and guidance

INTERVENTIONS:
Procedure: Advanced imaging for radiotherapy planning and guidance — Integration of MRI in the treatment planning process / Integration of daily cone-beam computed tomography (CBCT)

SUMMARY:
The integration of magnetic resonance imaging (MRI) in the treatment planning process for prostate cancer will reduce uncertainties in delineation of the prostate gland, and will enable delineation of the urethra, penile bulb, and internal pudendal artery. The integration of daily cone-beam computed tomography (CBCT) will markedly reduce set-up uncertainties, thereby reducing the minimum planning target volume (PTV) margin. By combining MRI simulation and daily CBCT, and by adapting radiation delivery accordingly, the investigators will reduce dose delivered to the rectum, bladder, urethra, and erectile structures. In this study, the investigators seek to determine whether this dose reduction translates to improved patient outcomes. In a prospective, 2-stage design, up to 190 patients will be enrolled. In the first stage, advanced imaging will be integrated without altering dose planning techniques. Stage 2 will reduce dose delivered to normal tissues, and will collect toxicity outcome measures. This clinical trial will be conducted over 3 years.

DETAILED DESCRIPTION:
Advances in medical imaging, and their integration in the treatment planning and daily guidance of radiotherapy, stand to improve the therapeutic ratio. Improved imaging can reduce uncertainties by 1) improving the accuracy and reproducibility of organ or tumor delineation, and 2) guiding and adapting delivery to account for organ motion. This paradigm has been widely accepted in the radiotherapy community, and much research has addressed the technical and dosimetric aspects for a sound clinical implementation. However, direct evidence of a clinical translation to improved patient outcomes is limited. In this study, we hypothesize that the integration of advanced imaging for treatment planning and guidance will safely enable a reduction of dose delivered to normal tissues, and will improve toxicity and quality of life (QOL) outcomes in patients receiving external beam radiotherapy for low or intermediate risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Low or intermediate risk localized prostate cancer:

* Gleason score ≤ 7
* PSA <20
* Stage T2a or less (Stage 2 only)
* <50% of biopsy cores involved with tumor (Stage 2 only)

Exclusion Criteria:

* History of hip replacement
* Inflammatory bowel disease or collagen vascular disease
* Contraindication to fiducial marker placement
* Bleeding diathesis or anticoagulant therapy that cannot safely be ceased temporarily
* Severe adverse event with prior TRUS-guided prostate biopsy
* Patient refuses fiducial marker placement
* Contraindication to MRI
* Patient randomization in PROFIT Trial (Stage 2 only)
* Patients not prescribed 78Gy in 39 fractions to the prostate gland.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-09; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To determine whether reducing the dose to normal tissues, enabled by the integration of advanced imaging, reduces the incidence of RTOG/CTC Grade ≥ 2 toxicity. | 10 years

SECONDARY OUTCOMES:
To determine whether reducing the dose to normal tissues, enabled by the integration of advanced imaging, improves quality of life in patients receiving external beam radiotherapy. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada